CLINICAL TRIAL: NCT06916000
Title: Effect of Ultrasound Guided Pericapsular Nerve Group (PENG) Block on Perioperative Pain Management in Patients Undergoing Hip Arthroplasty
Brief Title: Assessment of PENG Block as a Part of Multimodal Analgesia Following Hip Surgeries.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MS428/2024
Record Dates: First submitted 2024-11-28; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PENG block group (25 particiants) (Active Comparator): For postoperative pain management, all patients of this arm will receive 20 ml of 0.25% bupivcacaine according to the technique described by Giron-Arango.
  In addition, multimodal analgesia will be given including IV paracetamol 1000 mg BID and oral celecoxib tablet 100 mg BID. Also if needed nalbuphine 5 mg IV will be given as demand dose and when the NRS pain score was equal to or greater than 4 points.
  Interventions: Drug: Pericapsular nerve group (PENG) block
- Group C: control group (25 participants) (Experimental): Patients will receive only other multimodal analgesics
  Interventions: Other: Patients will receive only other multimodal analgesics including LCFN block via 10 ml of 0.25% bupivacaine.

INTERVENTIONS:
Drug: Pericapsular nerve group (PENG) block — As a part of multimodal analgesia patients will receive 20 ml of 0.25% bupivcacaine according to the technique described by Giron-Arango.
  All patients will receive the same analgesic protocol, which included IV paracetamol 1000 mg BID and NSAIDs if no contra-indication; PO celecoxib 100 mg BID. Also if needed nalbuphine 5 mg IV will be given as bolus demand dose and when the NRS pain score was equal to or greater than 4 points.
  Arms: PENG block group (25 particiants)
Other: Patients will receive only other multimodal analgesics including LCFN block via 10 ml of 0.25% bupivacaine. — Patients will receive only other multimodal analgesics including LCFN block via 10 ml of 0.25% bupivacaine.
  Arms: Group C: control group (25 participants)

SUMMARY:
to study the effect of Pericapsular nerve group (PENG) block as a part of multimodal analgesia regimen for hip arthroplasties

DETAILED DESCRIPTION:
PENG block is a novel block described by Giron-Arango in 2018 to anesthesize the anterior hip capsule as it is supplied by branches from femoral, obturator and accessory obturator nerves, sparing motor function is an additional significance So currently the block is used to reduce post operative opioid consumption, delay time rescue analgesia, facilitate positioning for spinal anesthesia for hip surgeries and to accelerate mobility and so hospital discharge saving this vulnerable group of patient from any hospital acquired pneumonia, decreasing hospital stays, and improving recovery times would provide valuable insights into its cost-effectiveness and long-term benefits for healthcare system Our primary outcome to be studied is pain assessment via Numer Rating Scale over 24 hours postoperatively, in addition to to secondary outcomes including the aforementioned advantages.

ELIGIBILITY:
Inclusion criteria:

* Age group: 18 years and older.
* ASA classification I to III.
* BMI : 18-35 .
* Gender: both sex

Exclusion criteria:

* Patient refusal.
* Patients on long-term pain medications.
* History of allergic reactions to local anesthetics
* Patients who had mental illness or uncooperative patients.
* BMI > 35 .
* Patients having coagulopathies or on anticoagulant or antiplatelet therapy.
* Severe cardiopulmonary disease
* ASA IV or more
* Diabetic or other neuropathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pain score: pain assessment using a Numeric Rating System (NRS) immediately in the postoperative period. | 24 hours
  Pain score: pain intensity will be evaluated using a Numeric Rating System (NRS) immediately in the postoperative period, every 2 hours during the first 6 hours and then every 6 hours till 24 hours postoperatively. Scores ranging from 0 to 10, with 0 indicating the absence of pain and 10 indicating the worst possible pain.

SECONDARY OUTCOMES:
Rescue analgesia timing and opioid consumption over 24 hours | 24 hours
  Time to first opioid demand and total opioid consumed by each patient individually over 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Ain Shams University, Abbasia, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No